CLINICAL TRIAL: NCT03994094
Title: Three Year Evaluation of a Cohort of Patients Presenting Osteoporotic Fractures
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2019-S7/01
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-06

CONDITIONS: Osteoporosis; Osteoporotic Fractures
MeSH Terms: conditions — Osteoporosis; Osteoporotic Fractures | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Telephone interview — Structured, directive, telephone interview, in order to collect the outcome measures in addition to the patients electronic health record.

SUMMARY:
A specialized osteoporosis clinic has existed in our hospital since 2010. The descriptive retrospective analysis of patients included in this pathway was the subject of a first study on patients included between January 2010 and January 2011 and reported to the Congress of the French Society of Rheumatology (SFR) in December 2011, then a second study on patients included between January 2012 and December 2016, presented as an e-poster at the SFR Congress in December 2017 and in a poster at the American Society of Bone and Mineral Research Conference (ASBMR) in October 2018 and published in 2019 in Archives of Osteoporosis.

The effectiveness specialized osteoporosis clinics is the subject of numerous publications.

It therefore seems important to evaluate the effectiveness of our management, 3 years from the date of inclusion of patients in the osteoporosis clinic of our hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had an osteoporotic fracture followed by the osteoporosis clinic since between January 2012 and December 2015
* Acceptation of the telephone interview

Exclusion Criteria:

* Age < 18 years
* No social security coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were enrolled in the cohort of the osteoporosis clinic of our hospital between january 2012 and December 2015 following an osteoporotic fracture.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Estimated)
Dates: Start 2019-06-12 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of fractures since the enrollment in the clinic | From the enrollment of patients between january 2012 and december 2015 to the interview date
  Number of incident fractures suffered by the patient since their enrollment in the osteoporosis clinic.

SECONDARY OUTCOMES:
Evolution of bone mineral density since the enrollment in the clinic | From the enrollment of patients between january 2012 and december 2015 to the interview date
  Evolution of the bone mineral density since their enrollment in the osteoporosis clinic
Satisfaction with the osteoporosis clinic | From the enrollment of patients between january 2012 and december 2015 to the interview date
  Level of satisfaction measured with a four level Lickert scale ( Very satisfied ? Satisfied? Unsatisfied? Dissatisfied?)

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte Haettich, MD, Principal Investigator — Centre Hospitalier du Mans, Rheumatology Department
Locations (1):
- Centre Hospitalier Le Mans, Le Mans, France

IPD SHARING:
Plan to Share IPD: No